CLINICAL TRIAL: NCT00067834
Title: Feasibility and Dosing Study of Bone Density Changes With and Without PEMF Following Immobilization of the Forearm
Brief Title: Electromagnetic Treatment For Bone Loss After Forearm Fracture
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N01 AR32267; NIAMS-091
Record Dates: First submitted 2003-08-28; First posted 2003-09-01 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Bone Disease, Metabolic; Osteopenia; Osteoporosis, Post-Traumatic
Keywords: Electromagnetic Fields; Bone; Forelimb; Radius
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis

INTERVENTIONS:
Device: Pulsing electromagnetic field (PEMF)

SUMMARY:
This study will determine the usefulness of pulsing electromagnetic field (PEMF) technology to reverse or reduce the bone loss (osteopenia) that occurs in the forearm after fracture or surgery.

DETAILED DESCRIPTION:
The long-range goal of this research is to develop a new and supplementary local treatment for osteoporosis to reduce the risk of fracture in susceptible individuals. PEMF is a noninvasive method to magnetically introduce a small amount of electrical current to a specific bone region to stimulate bone formation. PEMFs have been used for many years to treat nonunited fractures and enhance spine fusion healing and have been found to improve bone density in animal models of osteoporosis. Such a noninvasive intervention applied to the hip or spine, which are especially associated with high morbidity and mortality in aging individuals, could have a significant national health care impact.

If effective for the treatment of bone loss, PEMF technology may be effective in treating osteoporosis. The primary objective of this pilot study is to determine the feasibility of using PEMFs to reverse or reduce bone loss that occurs with disuse of the forearm after fracture or surgery and to determine the effect of daily treatment duration on efficacy.

Eighty patients who have recently undergone immobilization after hand surgery or after lower forearm fracture will be enrolled in this study. Participants will be randomized to either the PEMF group or a control group. PEMFs will be administered by means of a magnetic coil transducer placed over the treatment site for 1, 2, or 4 hrs/day for 8 weeks, beginning 6 weeks after the initial injury or surgery. A self-contained, battery-powered PEMF coil transducer already FDA-approved for fracture healing in the forearm will be used. Participants in the control group will receive inactive but otherwise identical units and treatment times. Measurements of bone density will be made using DEXA (dual energy x-ray absorptiometry) and pQCT (peripheral quantitative computer tomography) and compared to baseline. DEXA and pQCT provide planar and cross-sectional x-ray densitometry to determine forearm bone changes. Bone densities (global, cortical, and trabecular), bone cross-sectional structural geometry, and calculated strength index will be measured and compared to baseline values.

ELIGIBILITY:
Inclusion Criteria

* Treatment and immobilization for carpal instability or repair or a lower forearm fracture (Colles' or Smith's) within 6 weeks
* Intact, normal prior skeletal anatomy and function in both arms

Exclusion Criteria

* Previous forearm fracture (either arm), orthopedic procedure, or forearm deformity which might affect forearm bone density
* History of renal disease, liver disease, diabetes, hyperthyroidism, hyperparathyroidism, Cushing's disease, uncontrolled seizures, rheumatoid arthritis, Paget's disease, multiple myeloma, or hypothyroidism
* Implanted cardiac pacemakers or defibrillators
* Pregnant
* Drug therapies within the previous 3 months that could affect bone (e.g., bisphosphonates, estrogen, progesterone, CaF2, calcitonin, steroids, anti-seizure medications)
* Difficulties complying with the protocol due to physical or mental inability, drug or alcohol abuse, psychosis or dementia, imprisonment, or unavailable for follow-up
* History of osteoporosis, as defined by a DEXA T-score of more than 2 standard deviations below normal in the hip, spine, or unaffected forearm
* Prior osteoporotic hip or vertebral fracture

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2003-11; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Changes in bone density and geometry relative to baseline in the PEMF treated forearm during the 24 weeks after immobilization, as compared to the same changes in those receiving sham control treatment

SECONDARY OUTCOMES:
Changes in chemical markers of bone remodeling in the blood of PEMF treated versus sham control subjects
bone density and structural changes in the 24 weeks after immobilization, measured by comparing the treated versus the contralateral forearms in subjects receiving PEMF or sham treatment
influence of age, gender, and other factors

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A. Spadaro, PhD, Principal Investigator — Upstate Medical University Orthopedic Research Lab
Locations (1):
- Institute for Human Performance/Upstate Medical University, Syracuse, New York, United States